CLINICAL TRIAL: NCT00203697
Title: Minocycline Treatment in Patients With Idiopathic Pulmonary Fibrosis Being Treated With Standard of Care Therapy- a Pilot Study
Brief Title: Minocycline Therapy for Lung Scarring in Patients With Idiopathic Pulmonary Fibrosis - a Pilot Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-002Kleerup; NIH-NHLBI 1 P50 HL67665-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Eric Kleerup; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Minocycline

INTERVENTIONS:
Drug: minocycline

SUMMARY:
Pulmonary fibrosis is essentially scarring in the lungs. Some types (DIP, NSIP) most often respond to therapy. Others like UIP (usual interstitial pneumonitis) rarely respond. UIP frequently progresses and has a poor prognosis with a survival of three to five years. In UIP, most often the cause cannot be determined and is therefore called Idiopathic Pulmonary Fibrosis (IPF). A prevalence rate of 27-29 cases/100,000 has been reported that may even be as high as 250 cases/100,000 in individuals 75 years of age.

Idiopathic pulmonary fibrosis (IPF) is a chronic and fatal pulmonary disorder. Conventional treatment with immunosuppressive therapy has been disappointing, with a median survival of <40% at five years after diagnosis. Moreover, this therapy may lead to premature deaths that are a result of immunosuppression and susceptibility to infectious disease. Another problem related to IPF, is that we have an incomplete picture of the natural history of the pathogenesis of this disorder. Clearly, new strategies for therapy are necessary.

Published evidence suggests that less than 20% of patients with IPF respond to corticosteroids (prednisone). In patients that fail steroids, immunosuppressant drugs such as azathioprine or cyclophosphamide are used. An international consensus statement recommends both steroids and azathioprine or cyclophosphamide from the onset of treatment. Unfortunately a large number of trials have shown little or no effect of these drugs on the progression of disease. There are currently no FDA approved drugs for the treatment of IPF.

Laboratory findings establish that human specimens of Interstitial Lung Diseases including IPF demonstrate an impalance in expression of proteins (Th2 Cytokines, CC Chemokines, and CXC Chemokines). When these protein levels are in excess or low, they alter the normal lung mechanism, causing angiogenesis (abnormal blood vessel formation), inflammation, scar tissue formation and impaired immunity of the patient. We hope to establish that the efficacy of anti-angiogenetic agent as an add on therapy for IPF patients, will prove to bring stabilization or improvement.

Minocycline has been shown to inhibit angiogenesis (new abnormal blood vessel formation) and thus affect the fibrotic process (prevent scar tissue formation). Laboratory and animal studies support a potential therapeutic role for Minocycline in IPF.

Minocycline is a semi synthetic derivative of tetracycline. It was first marketed as an antibiotic in 1972. Clinical trials of minocycline have mainly been performed in sexually transmissible diseases and in acne. Minocycline is also used to treat several other diseases such as nocardiasis, mycobacteriosis, leprosy, lyme disease, pyoderma gangrenosum, autoimmune bullous dermatitis, carteaud disease, and prurigo. The usual side effects of minocycline are: lightheadedness, dizziness, or vertigo and pigmentation.

We will investigate genetic, molecular, cellular, whole animal models, and human specimens from patients with fibrotic lung disease to test our prediction: The pathogenesis of pulmonary fibrosis (lung scarring) is due to "multiple hits" that causes an inbalance of certain mediators (proteins) that are responsible for abnormal blood vessel formation, scar tissue formation (with and without inflammation inside the lungs) and impaired immunity of the patient. Each of the 3 projects in this proposal have a direct link to other projects and clinical core. The SCOR clinical core will identify and enroll patients with Interstitial Lung diseases (ILD), including IPF. The clinical core will collect clinical data, as well as obtain fluids from lung washings and human lung tissue specimens. Each project will use human specimens as indicated in each of their specific aims to correlate their findings with response to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical symptoms consistent with idiopathic pulmonary fibrosis (IPF) of > 3 months duration (insidious onset of otherwise unexplained dyspnea on exertion and bibasilar inspiratory crackles)
2. Age 20 through 79, inclusive. Patients ages 20-34 must have diagnosis by either open or video-assisted thoracoscopic (VATS) lung biopsy to be eligible.
3. Diagnosis must be made by high-resolution (HRCT) chest CT showing definite or probable IPF AND within 30 months prior to screening either of the following):

   * Open or VATS lung biopsy showing definite or probable usual interstitial pneumonia (UIP), required for subjects ages 20-34 due to the rarity of IPF in this age group OR
   * Non-diagnostic transbronchial biopsy to exclude other conditions (including granulomatous disease, sarcoidosis, hypersensitivity pneumonitis) AND
   * abnormal pulmonary function tests (reduced FVC or decreased DLCO or impaired gas exchange at rest or during exercise)

   AND 2 of the following:
   1. Age > 50 years
   2. Insidious onset of otherwise unexplained dyspnea on exertion
   3. Bibasilar, inspiratory crackles (dry or Velcro type in character)
4. Currently on low dose (< 0.3 mg/kg LBW) prednisone plus azathioprine or cyclophosphamide per ATS Consensus for at least 28 days prior to study treatment and intending to continue the same therapy until the end of study treatment. This therapy may be preceded by a course of higher-dose prednisone at the discretion of the treating physician.
5. FVC > 40% and < 90% of predicted (Hankinson/NHANES2) value at screening.
6. DLCO > 20% of predicted (Neas/NHANES3) value at screening.
7. PaO2 > 50 mmHg at rest after 20 minutes on room air at baseline.
8. Able to understand and sign a written informed consent form and comply with the requirements of the study.

Exclusion criteria

Patients with any of the following will be excluded from the study:

1. History of clinically significant environmental exposure known to cause pulmonary fibrosis (drugs, asbestos, beryllium, radiation, domestic birds, etc).
2. Known explanation for interstitial lung disease, other than IPF, including but not limited to radiation, sarcoidosis, hypersensitivity pneumonitis, bronchiolitis obliterans organizing pneumonia (BOOP), and cancer.
3. Diagnosis of any connective tissue disease (scleroderma, SLE, rheumatoid arthritis, etc.) according to the American College of Rheumatology criteria. Antinuclear antibody (UCLA test # 0737, $39) ≥1:160, rheumatoid factor (UCLA test #0881, $29) >25, Scl-70 positive (UCLA test #1977, $12), anticentromere antibodies positive (UCLA test #16232, $15) at baseline. These lab tests are considered minimum standard of care. Additional criteria, if evaluated (preferred standard of care) ENA (SM & RNP) (UCLA test number 16393, $36) positive and double strand DNA (UCLA test number 0797, $67) positive.
4. Any condition other than IPF, which in the opinion of the investigator, is likely to result in the death of the patient within the next year.
5. Evidence of active infection including bronchitis, sinusitis, UTI, cellulitis within 1 week prior to treatment.
6. History of unstable or deteriorating cardiac or neurologic disease, including but not limited to:

   1. Myocardial infarction, coronary artery bypass surgery or angioplasty within the past 6 months
   2. Congestive heart failure requiring hospitalization within the past 6 months
   3. Uncontrolled arrhythmia
   4. Stroke or TIAs within 18 months
7. Pregnant or lactating females. Females of child bearing potential are required to have a negative serum or urine pregnancy test prior to enrollment and agree to practice abstinence or prevent pregnancy by a medically acceptable method of birth control (e.g. barrier methods, IUD, Norplant, Provera injection or oral birth control pills).
8. Liver function above specific limits. Total bilirubin > 1.5 X ULN, transaminases (AST, SGOT) or (ALT, SGPT) > 3 ULN, alkaline phosphatase > 3 ULN.
9. Hematology outside of specified limits, WBC <2,500/mm3, hematocrit <30 or >59, platelets <100,000/mm3 at screening.
10. TSH outside the normal range (with or without thyroid supplementation at a stable dose for 3 months).
11. Investigational therapy for any indication within 28 days prior to treatment.
12. Investigational or clinical therapy including tetracycline (or derivatives), cyclosporin, methotrexate, chlorambucil, colchicine, d-penicillamine, pirfenidone, interferon-beta or interferon-gamma or other drugs (other than corticosteroids and azathioprine or cyclophosphamide) potentially affecting IPF within 6 months prior to treatment
13. Lung transplantation
14. Patients who would not be able to comply with the requirements for the trial.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kleerup, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Pulmonary Outpatient Clinic, Los Angeles, California, United States